CLINICAL TRIAL: NCT03449524
Title: Phase 2 Multicenter, Double-Blind, Placebo Controlled, Efficacy, Safety, and Pharmacokinetic Study of 2 Doses of CXA-10 on Stable Background Therapy in Subjects With Pulmonary Arterial Hypertension
Brief Title: PRIMEx - A Study of 2 Doses of Oral CXA-10 in Pulmonary Arterial Hypertension (PAH)
Acronym: PAH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: LOE
Sponsor: Complexa, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry); Philips Healthcare (Industry); Cardiovascular Clinical Sciences Inc (Industry); MicroConstants (Unknown); Innovative Analytics (Unknown); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CXA-10-301
Record Dates: First submitted 2018-02-14; First posted 2018-02-28 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: PAH
Keywords: Pulmonary Arterial Hypertension; Pulmonary Hypertension; PAH; Connective Tissue Disease-Associated; 6 Minute Walk Test; 6 Minute Walk Distance; Pulmonary Vascular Resistance; Cardiac MRI; Right Ventricular Function; Hypertension; Familial Primary Pulmonary Hypertension; Connective Tissue Diseases; Vascular Diseases; Cardiovascular Diseases; Hypertension, Pulmonary; Lung Diseases
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Hypertension; Familial Primary Pulmonary Hypertension; Connective Tissue Diseases; Vascular Diseases; Cardiovascular Diseases; Lung Diseases | interventions — CXA-10

STUDY DESIGN:
Intervention Model Description: CXA-10
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 75mg CXA-10 (Active Comparator): Once daily dosing of 75mg CXA-10 in the morning
  Interventions: Drug: 75mg CXA-10
- 150mg CXA-10 (Active Comparator): Once daily dosing of 150mg CXA-10 in the morning
  Interventions: Drug: 150mg CXA-10
- Placebo (Placebo Comparator): Once daily dosing in the morning
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 75mg CXA-10 — CXA-10 (10-nitro-9(E)-octadec-9-enoic acid) is a specific isomer of nitro-oleic acid (OA-NO2)
  Arms: 75mg CXA-10
Drug: 150mg CXA-10 — CXA-10 (10-nitro-9(E)-octadec-9-enoic acid) is a specific isomer of nitro-oleic acid (OA-NO2)
  Arms: 150mg CXA-10
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter double-blind, placebo-controlled study to evaluate the safety, efficacy and pharmacokinetics of 2 doses of CXA-10 on stable background therapy in 96 subjects 18 to 80 years of age with PAH.

DETAILED DESCRIPTION:
This is a multicenter double-blind, placebo-controlled study to evaluate the safety, efficacy and pharmacokinetics of 2 doses of CXA-10 on stable background therapy in 96 subjects 18 to 80 years of age with PAH.

The study will be performed in approximately 50 study centers across the United States of America and Europe. The recruitment period is anticipated to be approximately 24 months. Approximately 115 subjects will be enrolled to ensure at least 96 subjects complete the study.

Study participation for each subject will last approximately 8 months. The study will consist of a screening period (within 30 days prior to dosing), 180 days (approximately 6 months) treatment period and approximately 14 days follow-up period after the end of treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 to 80 years of age inclusive at Screening
* Weight ≥40 kg
* Must have a diagnosis of WHO Group 1 PH
* Have a World Health Organization (WHO) Classification of Functional Status Class II or III of patients with PH
* Must meet hemodynamic criteria by means of a right heart catheterization
* Meet pulmonary function test parameters
* A 6 MWD test of ≥125m and ≤550m at the visit
* Subjects must have a resting arterial oxygen saturation (SaO2) ≥90%, with or without supplemental oxygen, as measured by pulse oximetry at Screening
* Subjects enrolled in a prescribed exercise program for pulmonary rehabilitation must be in a stable program for 3 months prior to Screening (Visit 1) and must agree to maintain their current level of rehabilitation throughout the study. If subjects are not enrolled in a prescribed exercise training program for pulmonary rehabilitation, they cannot enroll during the Screening/Baseline Period or throughout the study
* If receiving simvastatin-containing products: dose should not exceed 20 mg/day
* Subjects must be receiving no more than three of the following previously approved PAH therapies: phosphodiesterase type 5 (PDE-5) inhibitors, endothelin receptor antagonist (ERA), soluble guanylate cyclase (sGC) stimulator, prostanoids, prostacyclin receptor agonists and must be on stable doses (≥3 months) at Screening (Visit 1)

Exclusion Criteria:

* Contraindications for CMRI imaging
* WHO Groups 2, 3, 4 and 5 Pulmonary Hypertension
* Unrepaired congenital heart defects and significant congenital heart defects (i.e., atrial septal defects, ventricular septal defects, and patent ductus arteriosus) repaired less than 1 year prior to Screening (Visit 1) (Group 1 classification of Pulmonary Hypertension)
* QTcF > 500 msec
* Acute myocardial infarction or acute coronary syndrome within the last 90 days
* Cerebrovascular accident/transient ischemic attack (CVA/TIA) within the last 90 days
* Hospitalization for left heart failure within the last 90 days
* Clinically significant aortic or mitral valve disease defined as greater than mild regurgitation or mild stenosis; pericardial constriction; restrictive or constrictive cardiomyopathy; left ventricular dysfunction (LVEF < 50%); left ventricular outflow obstruction; symptomatic coronary artery disease; autonomic hypotension; or fluid depletion
* Chronic atrial fibrillation and life-threatening cardiac arrhythmias
* Personal or family history of congenital prolonged QTc syndrome or sudden or sudden unexpected death due to a cardiac reason
* Clinically significant anemia
* Severe hepatic impairment or active chronic hepatitis
* Receiving intravenous inotropes within 2 weeks prior to Screening
* History of angina pectoris or other condition that was treated with long or short acting nitrates <12 weeks of Screening
* Received prednisone doses >15mg/day or changes in immunosuppressive medications < 12 weeks prior to Screening (Visit 1)
* Recent (within 1 year) history of abusing alcohol or illicit drugs.
* History of any primary malignancy, with no evidence of disease for at least 5 years
* Treatment with any investigational drug or device within 30 days or 5 half-lives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Right Ventricular Ejection Fraction (RVEF) | 6 months
  • To determine the efficacy of oral doses of CXA-10 on stable background therapy administered for 6 months in subjects with PAH assessed by right ventricular ejection fraction (RVEF) as measured by Cardiac MRI
Pulmonary Vascular Resistance (PVR) | 6 months
  • To determine the efficacy of oral doses of CXA-10 on stable background therapy administered for 6 months in subjects with PAH assessed by pulmonary vascular resistance (PVR) as measured by right heart catheterization (RHC)

SECONDARY OUTCOMES:
6 Minute Walk Distance (6MWD) | 6 months
  To determine the efficacy of oral doses of CXA-10 on stable background therapy administered for 6 months in subjects with PAH assessed by 6 minute walk distance (6MWD)

CONTACTS AND LOCATIONS:
Overall Officials: Theo Danoff, MD, Study Director — Complexa, Inc.
Locations (46):
- United States (40):
  - University of Alabama, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California San Francisco, San Francisco, California
  - University of Colorado Health, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Washington Hospital (Medstar), Washington D.C., District of Columbia
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida Health, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - AdventHealth, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesotta, Minneapolis, Minnesota
  - Washington University and Barnes Jewish Hospital, St Louis, Missouri
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - NYU Langone Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Christ Hospital-Lindner Research Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Penn State M.S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbuilt University, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Texas Tech, El Paso, Texas
  - Houston Methodist, Houston, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Inova Medical Campus, Falls Church, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Froedert Medical College of Wisconsin, Milwaukee, Wisconsin
- United Kingdom (6):
  - Golden Jubilee National Hospital, Glasgow
  - Royal Free, London
  - Royal Brompton, London
  - Hammersmith Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided